CLINICAL TRIAL: NCT05841680
Title: A Single-Session Intervention for Families on Waitlists for Child Anxiety
Brief Title: A Single-Session Intervention for Families on Waitlists for Child Anxiety Treatment
Acronym: aSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-0040
Record Dates: First submitted 2023-02-24; First posted 2023-05-03 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): Participants complete pre, post, and follow-up questionnaires. They have the option to view the SSI module after completing follow-up questionnaires.
- Single Session Intervention Receivers (Active Comparator): Participants complete pre then receive the SSI module. Then they complete post and follow-up questionnaires.
  Interventions: Behavioral: SSI Module

INTERVENTIONS:
Behavioral: SSI Module — Single Session Intervention (SSI) module for youth with anxiety disorders and their parents. The SSI module will include psychoeducation on the cognitive behavioral conceptualization of anxiety, introduction to self-regulation strategies to manage physiological manifestations of anxiety, and cognitive restructuring of anxiogenic thoughts. The SSI module will also involve parents and present strategies on how parents can support their children in managing anxious feelings and thoughts.
  Arms: Single Session Intervention Receivers

SUMMARY:
Lengthy wait times to access treatment for youth anxiety disorders is a critical issue. To help address this issue, investigators will pursue the following aims in N = 65 families on waitlists for outpatient youth anxiety psychosocial treatment. Aim 1 Pilot Phase: Develop and pilot a single session intervention (SSI) tailored for families on waitlists for outpatient psychosocial treatment for youth anxiety disorders. Investigators will pilot the single session intervention (SSI) with N = 5 families and use cognitive response interviewing to obtain data from parents and children, ensuring the content is understandable and accessible. The SSI will include psychoeducation on the cognitive behavioral conceptualization of anxiety, introduction to self-regulation strategies to manage physiological manifestations of anxiety, and cognitive restructuring of anxiogenic thoughts. The SSI will also involve parents and present strategies on how parents can support their children in managing anxious feelings and thoughts. Investigators will refine the SSI based on these data. Following the Pilot Phase, investigators will enroll an additional N = 60 families and randomize them to either the SSI (n = 30) or waitlist control (n = 30). Aim 2 Test Phase Acceptability, and Satisfaction: Examine acceptability of the refined SSI, as well as satisfaction with the SSI. Investigators hypothesize that users will find the module to be acceptable and will report high satisfaction. Aim 3 Test Phase Anxiety Outcomes: Demonstrate reductions in youth anxiety symptom severity. Investigators hypothesize that anxiety symptom severity and impairment will be significantly lower among youth who receive the refined SSI relative to youth on waitlist control. The main risk or discomfort from this research is that participants might feel uncomfortable answering questions about their behavior and feelings. Another possible risk is breach of confidentiality that could identify a participant as having elevated levels of anxiety. The benefits of this SSI would include increasing accessibility and scalability of treatment for youth anxiety disorders. Overall, this study will provide critically needed data to advance resource efficient treatment options for youth anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 7 and 17 years
* Endorse clinically elevated anxiety symptoms on either parent or youth report, as indicated by a score > 25 on the Screen for Child Anxiety and Related Emotional Disorders-Child or Parent Versions (SCARED-C/P).

Exclusion Criteria:

* Parent report of past diagnosis of Autism Spectrum Disorder, Intellectual Disability, Bipolar Disorder, Tourette's Disorder, Psychotic Disorders, or Substance Use Disorders
* Show high likelihood of hurting themselves or others
* Not having access/connectivity needed for telehealth video conferencing to complete the module.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Coral Gables, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 59 children were enrolled in this trial. Only children were enrolled. Parents provided parental consent for their child to participate, but were not considered enrolled. These 59 children were assigned to one of two arms: Waitlist Control or Single Session Intervention. Data were collected on these children and are reported in the Results. Data correspond to Aim 2 Test Phase Acceptability and Aim 3 Test Phase Anxiety Outcomes. Aim 1 Pilot Phase did not include quantitative data collection.
Period: Overall Study
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control | Single Session Intervention Receivers | Total
Number analyzed (Participants) | 29 | 30 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 12 | 16 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 25 | 26 | 51
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 25 | 49
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 30 | 59
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version at Posttreatment
Description: Posttreatment parent rating of youth anxiety symptom severity over the past week. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 35 (14) | 30 (12)

2. Primary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version at Posttreatment
Description: Posttreatment child rating of youth anxiety symptom severity over the past week. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 33 (14) | 23 (12)

3. Primary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version at Follow up
Description: Follow up parent rating of youth anxiety symptom severity over the past 3 weeks. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 34 (13) | 26 (14)

4. Primary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version at Follow-Up
Description: Follow up child rating of youth anxiety symptom severity over the past 3 weeks. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 31 (14) | 23 (13)

5. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version at Pre
Description: Child rating of youth anxiety symptom severity over the past month. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 36 (13) | 36 (10)

6. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version at Pre
Description: Parent rating of youth anxiety symptom severity over the past month. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 34 (13) | 37 (13)

7. Secondary Outcome: Child Anxiety Impact Scale - Parent Version at Pre
Description: Brief parent-report measure of anxiety-related functional impairment over the past month. The name of the measure is the Child Anxiety Impact Scale-Parent Version (CAIS-P). The CAIS-P is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-P range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 28 (14) | 22 (15)

8. Secondary Outcome: Child Anxiety Impact Scale - Child Version at Pre
Description: Brief youth-report measure of anxiety-related functional impairment over the past month. The name of the measure is the Child Anxiety Impact Scale-Child/Adolescent Version (CAIS-C). The CAIS-C is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-C range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 24 (14.) | 19 (11)

9. Secondary Outcome: Child Anxiety Impact Scale - Parent Version at Posttreatment
Description: Brief parent-report measure of anxiety-related functional impairment over the past week. The name of the measure is the Child Anxiety Impact Scale-Parent Version (CAIS-P). The CAIS-P is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-P range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 27 (15) | 18 (14)

10. Secondary Outcome: Child Anxiety Impact Scale - Child Version at Posttreatment
Description: Brief youth-report measure of anxiety-related functional impairment over the past week. The name of the measure is the Child Anxiety Impact Scale-Child/Adolescent Version (CAIS-C). The CAIS-C is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-C range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 21 (12) | 17 (14)

11. Secondary Outcome: Child Anxiety Impact Scale - Parent Version at Follow Up
Description: Brief parent-report measure of anxiety-related functional impairment over the past 3 weeks. The name of the measure is the Child Anxiety Impact Scale-Parent Version (CAIS-P). The CAIS-P is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-P range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 25 (15) | 15 (13)

12. Secondary Outcome: Child Anxiety Impact Scale - Child Version at Follow Up
Description: Brief youth-report measure of anxiety-related functional impairment over the past 3 weeks. The name of the measure is the Child Anxiety Impact Scale-Child/Adolescent Version (CAIS-C). The CAIS-C is a parent rated measure of anxiety-related functional impairment. Total scores on the CAIS-C range from 0 to 81, with higher scores representing more functional impairment.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 18 (12) | 16 (14)

13. Secondary Outcome: Family Accommodation Scale Anxiety - Parent Version at Pre
Description: Parent-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past month. The name of the measure is the Family Accommodation Scale Anxiety - Parent Version (FASA-P). The FASA-P is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 15 (8) | 13 (8)

14. Secondary Outcome: Family Accommodation Scale Anxiety - Child Version at Pre
Description: Youth-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past month. The name of the measure is the Family Accommodation Scale Anxiety - Child Version (FASA-C). The FASA-C is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: first session at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 15 (6) | 14 (7)

15. Secondary Outcome: Family Accommodation Scale Anxiety - Parent Version at Posttreatment
Description: Parent-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past week. The name of the measure is the Family Accommodation Scale Anxiety - Parent Version (FASA-P). The FASA-P is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 14 (8) | 11 (8)

16. Secondary Outcome: Family Accommodation Scale Anxiety - Child Version at Posttreatment
Description: Youth-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past week. The name of the measure is the Family Accommodation Scale Anxiety - Child Version (FASA-C). The FASA-C is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 11 (7) | 9 (6)

17. Secondary Outcome: Family Accommodation Scale Anxiety - Parent Version at Follow Up
Description: Parent-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past 3 weeks. The name of the measure is the Family Accommodation Scale Anxiety - Parent Version (FASA-P). The FASA-P is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 14 (9) | 11 (7)

18. Secondary Outcome: Family Accommodation Scale Anxiety - Child Version at Follow Up
Description: Youth-report measure of the frequency with which parents participate in their child's anxiety-related behaviors (e.g., assisting avoidance, providing reassurance) and modification of family routines because of child anxiety over the past 3 weeks. The name of the measure is the Family Accommodation Scale Anxiety - Child Version (FASA-C). The FASA-C is a measure of parental accommodation. Total scores on the FASA-C range from 0 to 36, with higher scores representing more parental accommodation.
Time Frame: 4 weeks after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control | Single Session Intervention Receivers
Number analyzed (Participants) | 29 | 30
units on a scale | 11 (7) | 8 (6)

19. Secondary Outcome: Client Satisfaction Questionnaire - Parent Report at Posttreatment
Description: Parent report measure of consumer satisfaction with services received (e.g., "How would you rate the quality of the services you received?" and "If a friend were in need of similar help, would you recommend our program to him or her?"). The name of the measure is Client Satisfaction Questionnaire (CSQ-8). Total scores on the CSQ-8 range from 8 to 32, with higher scores representing more satisfaction with services received.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Session Intervention Receivers
Number analyzed (Participants) | 30
units on a scale | 29 (3)

20. Secondary Outcome: Client Satisfaction Questionnaire - Youth Report at Posttreatment
Description: Youth-report measure of consumer satisfaction with services received (e.g., "How would you rate the quality of the services you received?" and "If a friend were in need of similar help, would you recommend our program to him or her?"). The name of the measure is Client Satisfaction Questionnaire (CSQ-8). Total scores on the CSQ-8 range from 8 to 32, with higher scores representing more satisfaction with services received.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Session Intervention Receivers
Number analyzed (Participants) | 30
units on a scale | 29 (2)

21. Secondary Outcome: Program Feedback Scale - Parent Report
Description: Parent-report measure of perceived acceptability of a single session intervention (e.g. "I enjoyed the program"). The name of the measure is the Program Feedback Scale (PFS). Total scores on the PFS range from 0 to 35, with higher scores representing more acceptability.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Session Intervention Receivers
Number analyzed (Participants) | 30
units on a scale | 34 (2)

22. Secondary Outcome: Program Feedback Scale - Youth Report
Description: Youth-report measure of perceived acceptability of a single session intervention (e.g. "I enjoyed the program"). The name of the measure is the Program Feedback Scale (PFS). Total scores on the PFS range from 0 to 35, with higher scores representing more acceptability.
Time Frame: 1 week after first session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Session Intervention Receivers
Number analyzed (Participants) | 30
units on a scale | 29 (5)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Waitlist Control | Single Session Intervention Receivers
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT05841680/Prot_SAP_000.pdf